CLINICAL TRIAL: NCT04700709
Title: Evaluate the Efficacy and Safety of RaparoBell® Tablet Plus Calcineurin Inhibitors Compared With Mycophenolate Mofetil Plus Calcineurin Inhibitors in ABO Incompatible De Novo Living Kidney Transplant Recipients. [ART Study]
Brief Title: Efficacy and Safety of Sirolimus Plus CNI Compared With MMF Plus CNI in ABO-i Kidney Transplant Recipients.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B110_01KT2002
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Kidney Transplantation
Keywords: Kidney Transplantation; ABO incompatible; Sirolimus
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RaparoBell® Tablet (Experimental): ABO-i De novo Living Kidney transplant recipients will be randomized after Kidney transplant.
  Interventions: Drug: Sirolimus Tab.
- Mycophenolate Mofetil Tablet/Capsule (Active Comparator): ABO-i De novo Living Kidney transplant recipients will be randomized after Kidney transplant.
  Interventions: Drug: Mycophenolate Mofetil Cap./Tab.

INTERVENTIONS:
Drug: Sirolimus Tab. — Orally, once-daily in the morning - The first dose is administered within maximum 6mg/day according to the investigator's judgement, check the blood concentration of Sirolimus at each visit and adjust the dose to acheive the blood concentration maintaining at 3~8ng/ml.
  Other Names: RaparoBell® Tab.
  Arms: RaparoBell® Tablet
Drug: Mycophenolate Mofetil Cap./Tab. — Up to 1g BID(total 2g daily), PO
  Other Names: Myrept® Cap./Tab.
  Arms: Mycophenolate Mofetil Tablet/Capsule

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of RaparoBell® Tablet Plus Calcineurin Inhibitors Compared with Mycophenolate Mofetil Plus Calcineurin Inhibitors in ABO incompatible De Novo Living Kidney Transplant Recipients.

DETAILED DESCRIPTION:
This study is Multi-center, Open-label, Randomized Controlled Phase 4 Study to Evaluate the Efficacy and Safety of RaparoBell® Tablet Plus Calcineurin Inhibitors Compared with Mycophenolate Mofetil Plus Calcineurin Inhibitors in ABO incompatible De Novo Living Kidney Transplant Recipients.

ELIGIBILITY:
Inclusion Criteria:

[Time of Screening]

1. Patients who plan to be transplanted ABO incompatible living donor kidney or not past 35 days after kidney transplantation
2. More than the age of 19 years old
3. Agreement with written informed consent

[Time of Randomization]

1. Patients who have transplanted Kidney within 4 weeks(25 days to 35 days)
2. Patients who take CNI plus MMF after kidney transplantation

Exclusion Criteria:

[Time of Screening]

1. Patients who have transplanted non-kidney organs or have plan to be transplanted non-kidney organs
2. PRA > 50% before desenitization or positive results of DSA
3. Receive a kidney from a related donor who showed HLA identical
4. Positive in serology test(HIV, HBsAg, HCV) in recipients and/or donor
5. Allergic/hypersensitivity reaction in the history of Investigational drugs or additives
6. Women who are pregnant or breast feeding or not agree to the proper use of contraception during the trial
7. Patient has conversation impairment because of mental illness within 6months
8. Participated in other trial within 4 weeks
9. In investigator's judgement

[Time of Randomization]

1. Patients with acute rejection who have been clinically treated after kidney transplantation
2. At the time of Randomization

   * Treatment with active liver disease or Liver function test(T-bilirubin, AST, ALT)is over 3 times than upper normal limit
   * WBC< 2,500/mm^3, or platelet < 75,000/mm^3, or ANC < 1,300/mm^3
3. Patients who had plasmapheresis within 1 week
4. Patents who had a record of taking mTOR inhibitor before
5. In investigator's judgement

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of composite efficacy failure | Until 48 weeks after taking medicine
  Composite efficacy failure include biopsy-confired acute rejection, graft loss, death, or follow-up failure

SECONDARY OUTCOMES:
Incidence of composite efficacy failure | Until 24 weeks after taking medicine
  Composite efficacy failure include biopsy-confired acute rejection, graft loss, death, or follow-up failure
Incidence of biopsy-confirmed acute rejection | Until 24weeks and 48weeks after taking medicine
  Banff Criteria
The pathological results and time of occurrence and method of treatment, result of the treatment of acute rejection confirmed by biopsy | Until 24weeks and 48weeks after taking medicine
  Banff Criteria
Survival rate | Until 24weeks and 48weeks after taking medicine
  transplanted organ and patients
Function of Kidney | Until 24weeks and 48weeks after taking medicine
  eGFR using MDRD(Modification of Diet in Renal Disease) method
Incidence of CMV, BKV infection | Until 24weeks and 48weeks after taking medicine
  Incidence of CMV, BKV infection

CONTACTS AND LOCATIONS:
Overall Officials: Kyu Ha Huh, M.D, Ph.D, Study Chair — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No